CLINICAL TRIAL: NCT05148208
Title: The Effect of Intradialytic Supplementation of Creatine in Chronic Hemodialysis Patients: a Pilot Study
Brief Title: Intradialytic Creatine Supplementation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202100665
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Dialysis; Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Supplementation of water
  Interventions: Device: Creatine supplementation to dialysate
- Creatine 0.5 mM (Active Comparator): Supplementation of creatine dissolved in water to a final concentration of 0.5 mM of creatine in the dialysate
  Interventions: Device: Creatine supplementation to dialysate
- Creatine 1 mM (Active Comparator): Supplementation of creatine dissolved in water to a final concentration of 1 mM of creatine in the dialysate
  Interventions: Device: Creatine supplementation to dialysate
- Creatine 1.5 mM (Active Comparator): Supplementation of creatine dissolved in water to a final concentration of 1.5 mM of creatine in the dialysate
  Interventions: Device: Creatine supplementation to dialysate
- Creatine 2.0 mM (Active Comparator): Supplementation of creatine dissolved in water to a final concentration of 2 mM of creatine in the dialysate
  Interventions: Device: Creatine supplementation to dialysate

INTERVENTIONS:
Device: Creatine supplementation to dialysate — Creatine supplementation to dialysate

SUMMARY:
We perform a pilot study to investigate whether intra-dialytic creatine supplementation via the dialysate will result in higher intra-erythrocyte creatine concentrations. Secondary outcomes will include changes in muscle mass, muscle strength and cognition.

DETAILED DESCRIPTION:
Dialysis is a life-saving treatment, but unfortunately health-related quality of life (HRQoL) of dialysis patients is poor and mortality risks are high compared to the general population. Although several potentially modifiable (e.g. pre-dialysis care and nutritional status) and unmodifiable risk factors (e.g. age and genetics) for excess risk of mortality and poor HRQoL have been identified in dialysis-dependent patients with chronic kidney disease (CKD), there is great need for identification of new potentially modifiable risk factors. We hypothesize that creatine deficiency is such a modifiable risk factor, which underlies several important causes for impaired HRQoL hemodialysis patients, such as protein energy wasting (PEW), sarcopenia, fatigue, muscle weakness, depression, cognitive impairment, and increased susceptibility and a higher risk of an adverse course of infectious diseases. We propose that creatine supplementation is particularly important for patients with dialysis-dependent CKD because (1) endogenous synthesis of creatine in these patients is severely impaired due to the virtual absence of kidney function and, consequently, the virtual absence of the first enzymatic step required for endogenous absence of creatine from the amino acids arginine and glycine (2) unopposed losses of creatine to the dialysis fluid during dialysis sessions, and (3) inadequate intake of creatine due to advices towards a primary plant-based diet in these patients. All this comes on top of the normally existing continuous non-enzymatic conversion of approximately 1.6-1.7% of the endogenous creatine pool to creatinine, which necessitates continuous replenishment of creatine by the combination of endogenous synthesis and dietary intake to remain in steady-state. This is a novel understanding because until recently it was not recognized that kidney function is an important contributor to endogenous creatine synthesis, so that the capacity to of patients with dialysis-dependent CKD to maintain creatine homeostasis in the light of ongoing conversion of creatine into creatinine, additional unopposed losses of creatine to the dialysis fluid and an inadequate dietary intake is severely impaired. Patients with dialysis-dependent CKD could benefit from creatine supplementation by allowing for maintenance of their endogenous creatine pools, which would help them to sustain bodily functions which depend on creatine availability, including normal function of muscles, heart, the immune system and brain.

Based on these novel/ recent findings, we hypothesize that creatine, intradialytic creatine supplementation may help to maintain creatine homeostasis among dialysis-dependent chronic kidney disease patients, and consequently improve muscle status, nutritional status, neurocognitive status fatigue and HRQoL.

Objective: The primary objective of this pilot study is the feasibility of prolonged intra-dialytic creatine supplementation.

The secondary objectives of this pilot study are to study the safety of prolonged intra-dialytic creatine supplementation for dialysis patients and finding the optimal dosage to replenish the creatine pool, to this end we will step wisely increase creatine concentrations of the dialysis solution (in the range of 0.5 mM to a maximum of 2mM, with the latter reflecting the concentration that can be reached after an oral bolus of creatine).

The third objective is to obtain pilot data on the effect of intradialytic creatine supplementation on muscle status, nutritional status, neurocognitive status fatigue and HRQoL to allow for calculation of the power for a lager intervention study.

Study design: Block-randomized double-blind placebo-controlled pilot study in 16 hemodialysis patients (which will be divided into four groups (0.5mM, 1.0mM, 1.5mM, 2.0mM) each consisting of three patients receiving creatine and one receiving placebo). The total study duration is 8 weeks with 6 weeks of active treatment and 2 weeks of wash-out.

Study population: The study population comprises of a total of 16 adult (≥18 years) clinically stable patients with dialysis-dependent chronic kidney disease treated by conventional hemodialysis in the UMCG and the Dialysis Center Groningen Intervention: Creatine will be added to the dialysis fluid and will thus be continuously administered during the whole hemodialysis session. We will study the effect of four increasing dosages of creatine (3 out of 4 patients per block) or placebo (1 out of 4 patients per block) in four groups of four patients: 0.5mM, 1.0mM, 1.5mM, or 2.0mM of creatine. The patients will receive creatine supplementation or placebo (sterile water with the same composition as the dialysate) during each hemodialysis session during a total period of 6 weeks. Creatine-monohydrate, Creapure® "Pharma Quality" (not GMP), produced by AlzChem Trostberg, Germany will be used for preparation of a 50 mmol/L stock solution of creatine which will be added to the dialysis fluid to reach the projected dialysate concentrations.

Main study parameters/endpoints: The main parameters for the pilot study are the plasma creatine concentration and intra-erythrocytic creatine concentration of both pre- and post-hemodialysis samples. Intra-erythrocytic creatine concentration will be used as a non-invasive proxy for creatine tissue uptake. Secondary study parameters are hand grip strength as a measure of muscle strength, the combined interdialytic urinary and intradialytic dialysate excretion of creatinine as a measure of muscle mass, and bioelectrical impedance analysis (BIA) as a measure of body composition and nutritional status. Other study parameters are N-terminal pro-brain natriuretic peptide (NT-proBNP) as a cardiac function marker, high sensitivity troponin T (hs-TNT) as a cardiac ischaemia marker, C-reactive protein as an inflammation marker, self-reported physical health using the EQ-6D, SF36, and the DSI, fatigue using the CIS and cognitive functions using the CFQ.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: For this study, during each of study visits (baseline, week 3, week 6, and after a wash-out period of 2 weeks) patients will have to stay at the dialysis unit for 45 minutes longer than usual for their regular HD treatment. Besides arterial blood sampling (from the dialysis line) no venepunctures are necessary. For each study visit the total blood volume will not exceed 152 ml. Participants with a residual diuresis of ≥ 200 ml per 24h are asked to collect interdialytic urine. During the hemodialysis session, the complete dialysate volume will be collected in a tank. Dialysate is considered a 'waste product' and the collection of dialysate is no burden for the patient. Questionnaires can be filled in during the hemodialysis session. None of the health tests performed as part of this study cause physical discomfort. To minimize any risk of falling, physical tests are performed prior to the dialysis session and under the supervision of an investigator. We believe it is justified to perform the proposed study in order to elucidate the possible effects of intra-dialytic creatine supplementation on e.g. muscle status, nutritional status, neurocognitive status fatigue in hemodialysis patients. The finding of a beneficial effect will improve HRQoL and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Hemodialysis treatment in the UMCG or DCG;
* Dialysis vintage ≥2 months;
* Conventional hemodialysis, thrice weekly treatment with three to five hours per dialysis treatment;
* Hemoglobin at previous routine monthly assessment greater than or equal to 6.5 mmol/l;
* Signed informed consent.

Exclusion Criteria:

* Pregnancy;
* Presence of clinical signs of infection;
* Confirmed diagnosis of malignancies;
* Incapacity of the Dutch language;
* Inability to complete questionnaires;
* Short life expectancy;
* Kidney transplantation planned within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Intra-erythrocyte creatine concentration | 6 weeks
  Intra-erythrocyte creatine concentration assessed by liquid chromatography mass spectrometry

IPD SHARING:
Plan to Share IPD: No